CLINICAL TRIAL: NCT04894526
Title: The Effect of Alternating Energy Intake Compared to Regular Energy Intake on the Fat Content in the Blood After a Meal in Abdominally Obese Adults
Brief Title: Alternating Energy Intake and Blood Fat Content After a Meal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: METC 20-089
Record Dates: First submitted 2021-04-20; First posted 2021-05-20 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Abdominal Obesity; Postprandial Lipemia; Lipid Metabolism; Glucose Metabolism
Keywords: Alternating Energy Intake; Abdominal Obesity; Postprandial Lipemia; Lipid Metabolism; Glucose Metabolism
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternating energy intake schedule (Experimental): To alternate between caloric overconsumption and caloric underconsumption from day-to-day
  Interventions: Other: Alternating Energy Intake
- Regular energy intake schedule (Active Comparator): To consume the usual energy intake on a daily basis
  Interventions: Other: Regular Energy Intake

INTERVENTIONS:
Other: Alternating Energy Intake — To alternate between caloric overconsumption (130% of usual total energy needs) and caloric underconsumption (70% of usual total energy needs) on a daily basis for 6 days/week followed by one ad libitum day for 4 weeks.
  Arms: Alternating energy intake schedule
Other: Regular Energy Intake — To consume the usual energy intake (100% of total energy needs) on a daily basis for 6 days/week, also followed by one ad libitum day for 4 weeks.
  Arms: Regular energy intake schedule

SUMMARY:
Increasing evidence suggests that meal timing affects metabolic health. For example, intermittent fasting (IF) may have positive effects on plasma glucose and lipid levels, insulin sensitivity, and blood pressure. However, IF protocols often result in significant weight loss. Therefore, it is not clear to what extent these beneficial metabolic effects are due to IF or to weight loss. Although the effect of IF independent of weight loss has been studied, daily energy intake in those studies did not differ between the days. Therefore, the investigators aim to examine the effect of alternating energy intake - i.e. standardised day-to-day fluctuations in energy intake - on metabolic health independent of weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women as judged by study physician
* Abdominally obese males (waist circumference ≥ 102 cm) and females (waist circumference ≥ 88 cm)
* Aged between 18 - 75 years
* Stable bodyweight (weight gain or loss ≤ 3 kg in the past three months)
* Willingness to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit
* Women should be pre- or postmenopausal
* Sedentary (light exercise < 1 h per week) or moderately active (moderate exercise 1-2 h per week)
* Having a general practitioner
* Agreeing that the participant and general practitioner will be informed about medically relevant personal test results by a physician
* Willing to comply to study protocol during study
* Informed consent signed

Exclusion Criteria:

* Fasting plasma glucose ≥ 7 mmol/l
* Fasting serum triacylglycerol ≥ 4.5 mmol/l
* Fasting serum total cholesterol ≥ 8 mmol/l
* Blood pressure ≥ 160/100 mm Hg
* Current smoker, or smoking cessation < 12 months
* Drug abuse
* Alcohol abuse (≥ 21 alcohol consumptions per week)
* Use of medication known to affect blood pressure, serum lipid metabolism, or glucose metabolism
* Having a medical condition or history which might impact study measurements, to be judged by the study physician (e.g. myocardial infarction, angina, thrombosis, stroke, cancer, familiar hypercholesterolemia, liver or bowel disease or diabetes)
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Women who are perimenopausal, have an irregular menstrual cycle, or are pregnant
* Use of over-the-counter and prescribed medication, which may interfere with study measurements (to be judged by the principal investigator), e.g. weight loss medication
* Reported dietary habits: medically prescribed diets or slimming diets
* Reported participation in night shift work 2 weeks prior to screening and/or during the study. Night work is defined as working between midnight and 6.00 AM

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Triacylglycerol area under the curve (AUC) | 4 hours
  The 4-hour AUC for triacylglycerol after consumption of a standardised mixed meal

SECONDARY OUTCOMES:
Fasting glucose metabolism | Baseline, week 2, and twice in week 4
  Fasting glucose metabolism (includes e.g. glucose and insulin concentrations)
Fasting lipid metabolism | Baseline, week 2, and twice in week 4
  Fasting serum lipid and lipoprotein profile
Marker for postprandial lipid metabolism | 4 hour period after consumption of a standardised mixed meal
  Marker for lipid metabolism includes triacylglycerol and will be measured after consumption of a standardised mixed meal
Markers for postprandial glucose metabolism | 4 hour period after consumption of a standardised mixed meal
  Markers for glucose metabolism include insulin and glucose and will be measured after consumption of a standardised mixed meal
24-hour glucose levels | 24 hours
  The total area under the curve (tAUC) for 24-hour glucose as measured with a continuous glucose sensor
Day-time glucose levels | From 07:00 to 22:00 (15 hours)
  The tAUC for day-time glucose (07:00 - 22:00 h) as measured with a continuous glucose sensor
Night-time glucose levels | From 22:01 to 06:59 (8 hours and 58 min)
  The tAUC for night-time glucose (22:01 - 06:59 h) as measured with a continuous glucose sensor
Glucose levels after main meal consumption | 2 hours
  The tAUC for glucose during 2 hours after main meal consumption (breakfast, lunch and dinner) as measured with a continuous glucose sensor.
The mean amplitude of glycemic excursions (MAGE) | 24 hours
  MAGE as parameter for the assessment of glycemic variability.
Continuous overall net glycemic action (CONGA) | 1 hour, 2 hours, and 4 hours
  CONGA to assess intraday glucose variability within predetermined time windows -> 1-hour interval (CONGA-1), 2-hour interval (CONGA-2), and 4-hour interval (CONGA-4).

OTHER OUTCOMES:
High-Sensitivity C-Reactive Protein (hs-CRP) levels | Baseline, week 2, and twice in week 4
  Fasting hs-CRP as inflammatory marker
Blood pressure | Baseline, week 2, week 3, and twice in week 4
  Office systolic and diastolic blood pressure
Body weight | Baseline, week 2, week 3, and twice in week 4
  Body weight in kilograms
Height | Baseline, week 2, week 3, and twice in week 4
  Height in centimeters
Body Mass Index | Baseline, week 2, week 3, and twice in week 4
  Body weight and height will be combined to report BMI in kg/m^2
Waist circumference | Baseline, week 2, week 3, and twice in week 4
  Waist circumference in centimeters
Hip circumference | Baseline, week 2, week 3, and twice in week 4
  Hip circumference in centimeters
Waist to hip ratio | Baseline, week 2, week 3, and twice in week 4
  Waist and hip circumference will be used to report the waist to hip ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands